CLINICAL TRIAL: NCT02099162
Title: Yonsei OCT (Optical Coherence Tomography) Registry for Evaluation of Efficacy and Safety of Coronary Stenting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2008-0030
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: OCT; Coronary; Stenting
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: coronary stents — e.g. Sirolimus eluting stent, Paclitaxel-eluting stent, Zotarolimus-eluting stent, Everolimus-eluting stent, Biolimus eluting stent, EPC(endothelial progenitor cell) Capture stent, etc

SUMMARY:
Optical coherence tomography (OCT) has been recently studied for evaluation of coronary stenting. Because of high resolutions, several reports have shown that OCT is appropriate for evaluating neointimal tissue after coronary stent implantation. Also, the strut coverage and the characterization of neointimal tissue can be accurately evaluated. Furthermore, OCT-defined coverage of a stent strut was proposed to be related with clinical safety in drug-eluting stents-treated patients. Therefore, the investigators will evaluate the appropriateness of currently using coronary stents (e.g. Sirolimus eluting stent, Paclitaxel-eluting stent, Zotarolimus-eluting stent, Everolimus-eluting stent, Biolimus eluting stent, EPC(endothelial progenitor cell) Capture stent, etc) based on the findings of OCT. Additionally, the investigators will evaluate neointimal hyperplasia, malposition or strut coverage to decide the differences in the stent characteristics, the duration of antiplatelet use, and the differences according to the clinical presentations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary stents
2. Patients who will have coronary stents because of coronary artery stenosis

Exclusion Criteria:

1. Hemodynamically unstable patients
2. Ostial lesions that begin within 15 mm of the left main coronary artery
3. Lesions with diameter more than 4 mm
4. Patients with allergy to antiplatelet agent (asprin or clopidogrel)
5. Patients with hepatic dysfunction (Liver enzyme 3 times the upper limit of normal)
6. Pregnant and lactating patients
7. Patients with life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited our tertiary hostpital (Severance Cardiovascular Hospital) for coronary angiography (with coronary stents or planning for coronary stents)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
OCT findings (stented lesions, native vessels) | at index PCI, at follow-up coronary angiography (3, 6, 9 or 12 months and at the time clinically indicated)
Clinical outcomes | up to 10 years
  Death, Cardiac death, Stent thrombosis, Myocardial infarction, Target-lesion revascularization, Target-vessel revascularization
Comparison of OCT findings with physiologic findings | at index PCI, at follow-up coronary angiography (3, 6, 9 or 12 months and at the time clinically indicated)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seodaemun-gu, Shinchondong, Seoul, South Korea

REFERENCES:
- [Derived] Kim BG, Kachel M, Kim JS, Guagliumi G, Kim C, Kim IS, Lee YJ, Lee OH, Byun YS, Kim BO, Milewski K, Lee SJ, Hong SJ, Ahn CM, Shin DH, Kim BK, Ko YG, Choi D, Jang Y. Clinical Implications of Poststent Optical Coherence Tomographic Findings: Severe Malapposition and Cardiac Events. JACC Cardiovasc Imaging. 2022 Jan;15(1):126-137. doi: 10.1016/j.jcmg.2021.03.008. Epub 2021 May 19. PMID 34023255